CLINICAL TRIAL: NCT07288151
Title: MDMA-Assisted Massed Exposure Therapy for PTSD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jessica Maples-Keller, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025P012039; TP240376 (Other: DOD)
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: MDMA; 3,4-Methylenedioxymethamphetamine; Massed prolonged exposure therapy; Pos traumatic stress disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MDMA group (Experimental)
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine (MDMA); Behavioral: Massed Prolonged Exposure (PE)
- Standard of Care (Placebo Comparator)
  Interventions: Drug: Placebo; Behavioral: Massed Prolonged Exposure (PE)

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine (MDMA) — MDMA is a synthetic compound, commonly administered as MDMA hydrochloride (HCl).
  The drug will be administered in 100mg doses for a single session on Visit 2 out of 10- day study sessions over 2 weeks. MDMA is administered orally in capsule form and is taken under supervision in a controlled, therapeutic environment
  Other Names: MDMA
  Arms: MDMA group
Drug: Placebo — Placebos will visually match the 3 MDMA capsules (40mg, 40mg, and 20mg).
  Arms: Standard of Care
Behavioral: Massed Prolonged Exposure (PE) — Massed exposure therapy will be conducted for 11 sessions, 10 daily sessions and an additional therapy session during V2. They will consist of repeated exposures to trauma memories (imaginal exposure) consistent with the manualized protocol for massed exposure therapy.
  Also consistent with this treatment manual, participants will listen to imaginal exposures outside of PE sessions for "homework."

SUMMARY:
The goal of this clinical trial is to investigate the efficacy of 3,4-methylenedioxy-methamphetamine hydrochloride (MDMA) combined with Massed Prolonged Exposure (PE) therapy for the treatment of posttraumatic stress disorder (PTSD) in adult participants diagnosed with PTSD. This randomized, placebo-controlled trial will enroll 95 participants.

The main questions it aims to answer are:

* Does the combination of PE + MDMA lead to greater reduction in PTSD symptom severity from pre-treatment to one-month follow-up compared to PE + placebo?
* Does PE + MDMA improve response efficiency and durability of PTSD symptom improvement compared to PE + placebo?
* Does MDMA + PE enhance extinction retention and reduce amygdala threat reactivity, and are these changes associated with improved PTSD outcomes?

Participants will:

* Receive 10 sessions of Massed Prolonged Exposure therapy over two weeks
* Be administered either 100 mg of MDMA or a placebo at Visit 2
* Undergo blinded independent evaluator assessments using the Clinician-Administered PTSD Scale for DSM-5-R (CAPS-5-R) at the one-month posttreatment follow-up

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) affects many individuals, including military veterans and civilians exposed to trauma. While trauma-focused therapies like Prolonged Exposure (PE) are effective, many people do not fully recover, and current medications often have limited success.

This study will test whether combining PE therapy with a single dose of MDMA (a psychoactive drug) can improve PTSD treatment outcomes. Ninety-five participants with PTSD will be randomly assigned to receive either MDMA or a placebo during the second of ten PE therapy sessions, which are delivered over two weeks. Researchers will measure PTSD symptoms one month after treatment using a standardized interview.

The study will also explore how MDMA affects brain responses related to fear and emotional memory, which may help explain how it works. Early results from a pilot study suggest this combination may lead to large reductions in PTSD symptoms. This is the first clinical trial to formally test MDMA with PE therapy, and it may lead to new, more effective treatment options for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis as assessed by Clinician-Administered Posttraumatic Stress Scale for DSM-5 - Revised (CAPS-5-R).
* Able to speak and read English (due to standardization of outcome measures).
* Willing to sign a release for the investigators to communicate with their primary care or mental health providers if indicated.
* Able to swallow pills.
* Agree to have study visits video and/or audio recorded, including Experimental Session, assessments, and non-drug therapy sessions.
* Willing to provide a contact (relative, spouse, close friend, or another support person) who is willing and able to be contacted by the investigators.
* Agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If able to become pregnant, must have a negative pregnancy test before study entry, at study entry, and before the Medicine Session. Must agree to use adequate birth control for a month before the Medicine session and through 10 days after the Medicine Session.
* Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications before the Medicine Session, and not participating in any other interventional clinical trials during the duration of the study, are driven home or to a hotel after the Medicine Session, and commit to medication dosing, therapy, and study procedures

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have previously participated in a Multidisciplinary Association for Psychedelic Studies (MAPS) sponsored MDMA clinical trial.
* Have any current problem which, in the opinion of the investigator or study physician, might interfere with participation.
* Have hypersensitivity to any ingredient of the Investigational Medicinal Product (IMP).
* Upon review of medical or psychiatric history and psychiatric assessment, have any current or past diagnosis that would be considered a risk to participating in the study
* Requires ongoing psychiatric medication use with certain exceptions. Individuals may decide to taper psychiatric medications under the guidance of their local provider.
* Have a history of any medical condition that could make receiving MDMA dangerous because of increases in blood pressure and heart rate or any medical condition the study physician believes would pose a safety risk or interfere with the effects of the treatment. Any medical disorder judged by the investigator to significantly increase the risk of MDMA administration by any mechanism is exclusionary.
* Have any unstable medical condition that would interfere with participation.
* Have uncontrolled hypertension) documented on three separate occasions.
* Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
* Have a history of ever having ventricular arrhythmia or any other abnormal heart rhythm that the study physician believes would pose a significant risk of participation.
* Have an abnormal finding on electrocardiogram
* Have a history of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Require the use of concomitant medications that could impact the effects or safety of MDMA during the Medicine Session.
* Have symptomatic liver disease or significant liver enzyme elevations.
* Have a history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (105 lbs.).
* Are pregnant or nursing
* Have engaged in ketamine-assisted therapy or used ketamine within 12 weeks of enrollment

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD symptoms measured by CAPS-5-R | Baseline, 1 month post-treatment
  The CAPS-5-R is a structured clinical interview used to assess PTSD symptoms based on DSM-5 criteria. Each symptom is rated on frequency and intensity
  * Combined into a severity score per item
  * Total score reflects overall PTSD symptom severity

SECONDARY OUTCOMES:
Changes in PTSD symptoms measured by PCL-5 | Baseline, 1 month post treatment
  The PCL-5 is a 20-item self-report questionnaire used to measure PTSD symptoms based on DSM-5 criteria. Participants rate how much they've been bothered by each symptom in relation to a specific traumatic event, using a scale from 0 ("Not at all") to 4 ("Extremely"). A total score of 33 or higher indicates clinically elevated PTSD symptoms
Change in PHQ questionnaire scores | Baseline, 1 month post-treatment
  The PHQ-9 is a questionnaire used to assess depression severity. Each of the 9 items is scored from 0 to 3, giving a total score between 0 and 27.
  Higher scores suggest more severe depressive symptoms.

OTHER OUTCOMES:
Changes in fMRI-based neural activation patterns | Day 1 of treatment, Day 10 of treatment
  Participants will view 15 blocks of fearful face stimuli and 15 blocks of neutral face stimuli, with emotion condition randomly interweaved. Within each block, 8 face stimuli will be presented for 500 ms each, followed by a 500 ms intertrial interval.
  Changes in fMRI-based neural activation patterns following MDMA-assisted massed exposure therapy will be reported.
Changes in fear extinction retention | Day 4, Day 10 of treatment
  This will be assessed via a Pavlovian fear conditioning/extinction paradigm in which colored shapes are presented visually and paired with a 250 millisecond air blast.
  Changes in fear extinction retention following MDMA-assisted massed exposure therapy will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Maples-Keller, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Brain Health Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No